CLINICAL TRIAL: NCT01912352
Title: Gene-environment Interactions and Brain Functional Connectivity Associated With Norepinephrine System Genes in Attention Deficit Hyperactivity Disorder
Brief Title: Gene-environment Interactions and Brain Functional Connectivity in Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University (Other)
Collaborators: Korea Research Foundation (Other)
Responsible Party: Principal Investigator, Jae-Won Kim, Professor, Seoul National University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2010-0002283
Record Dates: First submitted 2013-07-16; First posted 2013-07-31 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-11

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; ADRA2A; Methylphenidate; Response
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Methylphenidate (Experimental): Participants were treated with methylphenidate (ranging from to 63mg) for 8 weeks. Doses of methylphenidate were titrated depending on symptoms and adverse eff ects at the 2nd and 4th weeks of treatment.
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate

SUMMARY:
The aims of the current study are to examine gene-environment interactions associated with norepinephrine (NE) system genes (ADRA2A, SLC6A2) in ADHD, and to evaluate whether genetic changes in norepinephrine pathway are associated with differences in functional connectivity of white matter fiber tracts, as measured by diffusion tensor imaging (DTI). Furthermore, this study aims to examine neurobiological markers, such as intermediate neuroimaging phenotypes or neuropsychological endophenotypes associated with the pathophysiology of ADHD. Through evaluating drug responses and side effects with the associated measures of clinical, neuropsychological and neuroimaging characteristics, investigators would like to investigate predictors of treatment response associated with NE system genes in ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Attention-deficit Hyperactivity Disorder
* 6-18 years old

Exclusion Criteria:

* History of neurological diseases, including convulsive disorders or brain damage
* IQ below 70
* Pervasive developmental disorder (autism)
* Language difficulties or learning disorders (reading disorders, mathematics disorders and disorders of written expression).
* Tourette's syndrome
* Bipolar disorder
* Psychosis

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2010-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Won Kim, MD., PhD., Principal Investigator — Seoul National University and Seoul National University Hospital

REFERENCES:
- [Derived] Kim JI, Kim JW, Shin I, Kim BN. Effects of Interaction Between DRD4 Methylation and Prenatal Maternal Stress on Methylphenidate-Induced Changes in Continuous Performance Test Performance in Youth with Attention-Deficit/Hyperactivity Disorder. J Child Adolesc Psychopharmacol. 2018 Oct;28(8):562-570. doi: 10.1089/cap.2018.0054. Epub 2018 Jun 15. PMID 29905488
- [Derived] Kim JW, Sharma V, Ryan ND. Predicting Methylphenidate Response in ADHD Using Machine Learning Approaches. Int J Neuropsychopharmacol. 2015 May 10;18(11):pyv052. doi: 10.1093/ijnp/pyv052. PMID 25964505
- [Derived] Hong SB, Zalesky A, Park S, Yang YH, Park MH, Kim B, Song IC, Sohn CH, Shin MS, Kim BN, Cho SC, Kim JW. COMT genotype affects brain white matter pathways in attention-deficit/hyperactivity disorder. Hum Brain Mapp. 2015 Jan;36(1):367-77. doi: 10.1002/hbm.22634. Epub 2014 Sep 9. PMID 25201318

RESULTS

PARTICIPANT FLOW:
Groups:
- Methylphenidate: Participants were treated with methylphenidate (raning from 10mg to 63mg) for 8 weeks. Doses of MPH were titrated depending on symptoms and adverse eff ects at the 2nd and 4 th weeks of treatment.
Period: Overall Study
Arm/Group | Methylphenidate
Started | 83
Completed | 78
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Methylphenidate
Number analyzed (Participants) | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.5 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 65
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 83
Scores on the ADHD Rating Scale-IV [Mean (Standard Deviation); unit: units on a scale] — Attendtion-deficit hyperactivity disorder (ADHD) Rating Scale-IV is the sum of 18 questions, ranging from 0 (no symptoms) to 54 (worst possible symptoms).
  units on a scale | 26.1 (10.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline ADHD Rating Scale-IV Scores at 8 Weeks
Description: Attendtion-deficit hyperactivity disorder (ADHD) Rating Scale-IV is the sum of 18 questions, ranging from 0 (no symptoms) to 54 (worst possible symptoms).
  Change from baseline ADHD Rating Scale-IV scores at 8 weeks was calculated as baseline minus 8 weeks.
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate
Number analyzed (Participants) | 78
units on a scale | 14.9 (10.9)

2. Secondary Outcome: Clinical Global Impression-Improvement Scale at 8 Weeks
Description: Clinical Global Impression-Improvement (CGI-I) scale is a one-item measure evaluating the change from the initiation of treatment on a seven-point scale: "Compared to the patient's condition at baseline [prior to medication initiation], this patient's condition is: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment.
  Clinical Global Impression-Improvement was measured at 8 weeks.
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate
Number analyzed (Participants) | 78
units on a scale | 2.3 (0.7)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Methylphenidate
Serious Adverse Events (participants affected / at risk) | 0/83
Other Adverse Events (participants affected / at risk) | 47/83
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methylphenidate (N=83)
Headache (Nervous system disorders) | 1
decreased appetite (Gastrointestinal disorders) | 36
stomach pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Tiredness (Nervous system disorders) | 1
Irritability (Psychiatric disorders) | 3
Trouble sleeping (Psychiatric disorders) | 9
Nail biting (Psychiatric disorders) | 2
Proness to crying (Psychiatric disorders) | 1
Tic (Psychiatric disorders) | 1
Depressive mood (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Excitability (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No